CLINICAL TRIAL: NCT00884533
Title: A Study to Evaluate the Effect of Extended Release Rosiglitazone (RSG XR) on Cardiac Conduction as Compared to Placebo and a Single Oral Dose of Moxifloxacin
Brief Title: QTc Study of Rosi XR in Healthy Volunteers
Acronym: Rosi XR
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The whole project was terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111802
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer's Disease
Keywords: QTc; pharmacokinetics; rosiglitazone XR; cardiac conduction; healthy volunteers
MeSH Terms: conditions — Alzheimer Disease | interventions — Moxifloxacin

ARMS (3):
- Group 1 (Experimental): Group 1 - placebo on Day -1, rosi XR 8mg from Days 1-20, rosi XR 20mg on Day 21
  Interventions: Drug: Rosi XR; Other: Placebo
- Group 3 (Placebo Comparator): Placebo on Day -1, Days 1-20 and Day 21
  Interventions: Other: Placebo
- Group 2 (Active Comparator): Placebo for Day -1, placebo on Days 1-20 and moxifloxacin active comparator 400 mg on Day 21
  Interventions: Other: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Rosi XR — Rosi XR
  Arms: Group 1
Other: Placebo — Placebo
Drug: Moxifloxacin — 400mg single dose
  Arms: Group 2

SUMMARY:
This study is a randomised double blind, parallel group, and will evaluate the effects of repeat oral doses of RSG- XR for 21 days on the QTc interval compared to placebo in a population of healthy adult males and females.

DETAILED DESCRIPTION:
An extended release (XR) formulation of rosiglitazone maleate (RSG), a new formulation of rosiglitazone, is being investigated as a treatment for patients with mild to moderate Alzheimer's disease (AD).

This study is a randomised double blind, parallel group, and will evaluate the effects of repeat oral doses of RSG- XR for 21 days (due to the long half-life of the main metabolite M10) on the QTc interval compared to placebo in a population of healthy adult males and females between 18 and 45 years of age. Moxifloxacin, a drug with well-quantified QTc prolongation, will be included as a positive control in order to validate the ability of the study to detect small changes in QTc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 18 and 45
* Female of non child bearing potential or if of child bearing potential they must use adequate contraception for the duration of the study up until 14 days after the last dose
* Body weight greater than or equal to 45 kg and BMI within the range 19 - 32 inclusive
* Subjects must provide full written informed consent

Exclusion Criteria:

* Cardiac conduction abnormalities
* Any history of myocardial infarction, syncope, or cardiac arrhythmias or a history of uncontrolled hypertension or unstable heart disease
* Subjects with a systolic blood pressure outside the range of 90 to 150 mmHg or diastolic blood pressure outside the range of 50 to 100 mmHg
* Subjects with a personal or family history of QTc prolongation or unexplained cardiac arrest.
* Has a history of illicit drug use or alcohol abuse within the past year or a positive pre-study test for alcohol, cotinine, or drugs of abuse at Screening or prior to the start of dosing
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase values greater than 2.5 times the ULN, total bilirubin values >1.5 times the upper limit of normal (ULN), or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C)
* A positive test at Screening for Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV)
* Use of any agents that are known to inhibit or induce cytochrome CYP3A4 enzymes within 7 days prior to the first dose of study drug (including foods or supplements such as grapefruit-containing products, mustard greens, kale, kohlrabi, broccoli, collard greens, brussel sprouts, watercress, charbroiled meats or St. John's Wort
* Use of any prescription or non-prescription drugs, in particular drugs known to inhibit or induce CYP2C8, vitamins (exceptions may be considered on a case-by-case basis with the GSK medical monitor), herbal and dietary supplements within fourteen days prior to the first dose of study drug
* Lactating or pregnant females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Day 20 time-matched change from baseline in QTcI for RSG- XR 8mg and placebo | Day 20
Day 21 time-matched change from baseline in QTcI for RSG- XR 20mg, placebo and moxifloxacin 400mg | Day 21

SECONDARY OUTCOMES:
Day 20 time-matched change from baseline in QTcF and QTcB for RSG XR 8mg and placebo. | Day 20
Day 21 time-matched change from baseline in QTcF and QTcB for RSG XR 20mg, placebo and moxifloxacin 400mg | Day 21
Tolerability of repeat doses of RSG- XR at 8 mg and a single oral dose of RSG- XR at 20 mg as assessed by 12-lead ECGs, vital signs, adverse events, and clinical laboratory tests. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Overland Park, Kansas, United States
- GSK Investigational Site, London, United Kingdom